CLINICAL TRIAL: NCT01050556
Title: Folic Acid and Creatine as Therapeutic Approaches for Lowering Blood Arsenic
Acronym: FACTA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mary Gamble, Associate Professor of Environmental Health Sciences, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AAAC8618; R01CA133595 (NIH)
Record Dates: First submitted 2010-01-13; First posted 2010-01-15 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: High Blood Arsenic Due to Chronic Arsenic Exposure
Keywords: arsenic; folate; folic acid; creatine; arsenicosis; nutrition
MeSH Terms: interventions — Folic Acid; Creatine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Placebo (Placebo Comparator): Placebo daily
  Interventions: Other: Placebo
- Folic Acid 400 ug (Experimental): 400 µg folic acid daily
  Interventions: Dietary Supplement: folic acid
- Folic Acid 800 ug (Experimental): 800 µg folic acid daily
  Interventions: Dietary Supplement: folic acid
- Creatine (Experimental): creatine daily
  Interventions: Dietary Supplement: creatine
- Creatine + Folic Acid (Experimental): creatine + folic acid daily
  Interventions: Dietary Supplement: creatine + folic acid

INTERVENTIONS:
Other: Placebo — daily, 24 weeks
  Arms: Placebo
Dietary Supplement: folic acid — 400 ug/d for 12 or 24 weeks
  Arms: Folic Acid 400 ug
Dietary Supplement: folic acid — 800 µg/d for 12 or 24 weeks
  Arms: Folic Acid 800 ug
Dietary Supplement: creatine — 3 mg/d for 12 weeks
  Arms: Creatine
Dietary Supplement: creatine + folic acid — 3 mg creatine/d + 400 µg folic acid/d for 12 weeks
  Arms: Creatine + Folic Acid

SUMMARY:
The purpose of this study is to determine whether folic acid, alone or together with creatine supplementation, can lower blood arsenic concentrations and improve the ability to detoxify arsenic.

DETAILED DESCRIPTION:
Approximately 140 million people in over 70 countries are chronically exposed to arsenic (As)-contaminated drinking water at concentrations far exceeding the World Health Organization standard of 10 µg/L. As is a carcinogen known to cause cancers of the skin, bladder, and lung, as well as ischemic heart disease and neurologic impairments. Methylation of ingested inorganic arsenic (InAs) to methylarsonic-(MMA) and dimethylarsinic acids (DMA) relies on folate-dependent one carbon metabolism, utilizing S-adenosylmethionine (SAM) as the methyl donor, and facilitates urinary As elimination. The results from our Nutritional Influences on Arsenic Toxicity (NIAT) study indicate that folate deficiency and hyperhomocysteinemia (HHcys) are associated with a reduced capacity to methylate arsenic and are risk factors for arsenic-induced skin lesions. Furthermore, folic acid (FA) supplementation does indeed facilitate As elimination and significantly lowers blood As concentrations in individuals who are folate deficient. We have also determined that blood As is a good biomarker of As exposure and is directly associated with the risk for As-induced skin lesions. Collectively, the implication of these findings is that FA has enormous therapeutic potential for ameliorating the long-term health consequences of arsenic exposure for the many populations at risk. However, several fundamental questions remain and will be addressed in this study. This trial is designed to determine 1) whether FA supplementation lowers blood As concentrations in the general Bangladeshi population, 2) at what time point a nadir in blood As is achieved, and 3) whether creatine supplementation, alone or in addition to 400 µg/d FA, will spare methyl groups, resulting in lower blood As, lower homocysteine (Hcys) concentrations, and increased methylation of As. The creatine arms are based on multiple studies that show that urinary creatinine concentrations are a very strong predictor of As methylation. The final step in creatine biosynthesis is the methylation of guanidinoacetate to creatine; this process consumes 50-75% of all SAM-derived methyl groups and is also responsible for 50-75% of all Hcys biosynthesis. Thus, this trial will test the hypothesis that creatine supplementation, which shuts down endogenous creatine biosynthesis, will spare methyl groups, lower Hcys, and increase As methylation.

ELIGIBILITY:
Inclusion Criteria:

* Currently exposed to arsenic via contaminated drinking water
* Well water arsenic concentration > 10 ug/L
* Between the ages of 20 and 65

Exclusion Criteria:

* Women who are currently pregnant or plan to become pregnant within the next 6 months
* Currently taking nutritional supplements
* Known renal disease
* Participation in any other clinical trial

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2010-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
blood arsenic concentrations | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mary V Gamble, PhD, Principal Investigator — Columbia University, Department of Environmental Health Sciences
Locations (1):
- Columbia University Arsenic Research Project, Dhaka, Bangladesh

REFERENCES:
- [Derived] Li W, Wu H, Goldsmith J, Glabonjat RA, Ilievski V, Balac O, Slavkovich V, Pinto-Pacheco B, Lin X, Parvez F, Jackson GL, Siddique AB, Uddin MN, Islam T, Martinez-Morata I, Navas-Acien A, Niedzwiecki MM, Kioumourtzoglou MA, Pierce BL, Graziano JH, Bottiglieri T, Walker DI, Gamble MV. Metabolic Signature of Arsenic Exposure and Metabolism: The Folic Acid and Creatine Trial. Environ Sci Technol. 2025 Jul 29;59(29):14905-14916. doi: 10.1021/acs.est.5c01597. Epub 2025 Jul 16. PMID 40668877
- [Derived] Martinez-Morata I, Wu H, Galvez-Fernandez M, Ilievski V, Bottiglieri T, Niedzwiecki MM, Goldsmith J, Jones DP, Kioumourtzoglou MA, Pierce B, Walker DI, Gamble MV. Metabolomic Effects of Folic Acid Supplementation in Adults: Evidence from the FACT Trial. J Nutr. 2024 Feb;154(2):670-679. doi: 10.1016/j.tjnut.2023.12.010. Epub 2023 Dec 12. PMID 38092151
- [Derived] Abuawad AK, Bozack AK, Navas-Acien A, Goldsmith J, Liu X, Hall MN, Ilievski V, Lomax-Luu AM, Parvez F, Shahriar H, Uddin MN, Islam T, Graziano JH, Gamble MV. The Folic Acid and Creatine Trial: Treatment Effects of Supplementation on Arsenic Methylation Indices and Metabolite Concentrations in Blood in a Bangladeshi Population. Environ Health Perspect. 2023 Mar;131(3):37015. doi: 10.1289/EHP11270. Epub 2023 Mar 28. PMID 36976258
- [Derived] Bae S, Kamynina E, Guetterman HM, Farinola AF, Caudill MA, Berry RJ, Cassano PA, Stover PJ. Provision of folic acid for reducing arsenic toxicity in arsenic-exposed children and adults. Cochrane Database Syst Rev. 2021 Oct 18;10(10):CD012649. doi: 10.1002/14651858.CD012649.pub2. PMID 34661903
- [Derived] Bozack AK, Howe CG, Hall MN, Liu X, Slavkovich V, Ilievski V, Lomax-Luu AM, Parvez F, Siddique AB, Shahriar H, Uddin MN, Islam T, Graziano JH, Gamble MV. Betaine and choline status modify the effects of folic acid and creatine supplementation on arsenic methylation in a randomized controlled trial of Bangladeshi adults. Eur J Nutr. 2021 Jun;60(4):1921-1934. doi: 10.1007/s00394-020-02377-z. Epub 2020 Sep 11. PMID 32918135
- [Derived] Bozack AK, Hall MN, Liu X, Ilievski V, Lomax-Luu AM, Parvez F, Siddique AB, Shahriar H, Uddin MN, Islam T, Graziano JH, Gamble MV. Folic acid supplementation enhances arsenic methylation: results from a folic acid and creatine supplementation randomized controlled trial in Bangladesh. Am J Clin Nutr. 2019 Feb 1;109(2):380-391. doi: 10.1093/ajcn/nqy148. PMID 30590411
- [Derived] Hall MN, Howe CG, Liu X, Caudill MA, Malysheva O, Ilievski V, Lomax-Luu AM, Parvez F, Siddique AB, Shahriar H, Uddin MN, Islam T, Graziano JH, Gamble MV. Supplementation with Folic Acid, but Not Creatine, Increases Plasma Betaine, Decreases Plasma Dimethylglycine, and Prevents a Decrease in Plasma Choline in Arsenic-Exposed Bangladeshi Adults. J Nutr. 2016 May;146(5):1062-7. doi: 10.3945/jn.115.227132. Epub 2016 Apr 6. PMID 27052531
- [Derived] Peters BA, Hall MN, Liu X, Parvez F, Siddique AB, Shahriar H, Uddin MN, Islam T, Ilievski V, Graziano JH, Gamble MV. Low-Dose Creatine Supplementation Lowers Plasma Guanidinoacetate, but Not Plasma Homocysteine, in a Double-Blind, Randomized, Placebo-Controlled Trial. J Nutr. 2015 Oct;145(10):2245-52. doi: 10.3945/jn.115.216739. Epub 2015 Aug 26. PMID 26311810